CLINICAL TRIAL: NCT04993833
Title: Inter-Device Reliability of the NPi-300 Pupillometer
Acronym: TRIPLE
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: NeurOptics Inc. (Industry)
Responsible Party: Principal Investigator, DaiWai Olson, Director of Neuroscience Nursing Research Center, University of Texas Southwestern Medical Center
Other Study IDs: STU-2021-0693
Record Dates: First submitted 2021-07-13; First posted 2021-08-06 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Critical Illness; Neuropathy
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Patients: Patients with risk of cerebral edema.
  Interventions: Device: NPi-200 and NPi-300 pupillometers
- Healthy Control: Staff/Faculty who interact with patients at the enrolling site.
  Interventions: Device: NPi-200 and NPi-300 pupillometers

INTERVENTIONS:
Device: NPi-200 and NPi-300 pupillometers — Device which measures PLR.

SUMMARY:
The purpose of this study is to explore the inter-device reliability between the NPi-200 and NPi-300.

DETAILED DESCRIPTION:
Paired assessments will be made on patients who are consented; and on healthy controls who have verbally assented to participate. We plan to enroll 20 patients and 50 healthy controls. Assessments will be made at the convenience of the patient and healthy controls. Each assessment will include bilateral PLR reading within a 5 minute interval. The first assessment will be completed with the NPi-200 and the second assessment will use the NPi-300. The data will be entered into a CRF.

If there is a significant difference between readings from the NPi-200 and the NPi-300, we will repeat the bilateral assessment in the following hour and the regularly scheduled time.

ELIGIBILITY:
Inclusion Criteria (Patient Cohort):

* Subjects will be included if they are adults (>18 years of age) and have a neurological or neurosurgical diagnosis that place them at risk for cerebral edema. Subjects also have to be admitted to the enrolling site. Persons consenting for the study (whether patient or LAR) will need to be able to consent for the study in English.

Exclusion Criteria (Patient Cohort):

* Patients that will be excluded from the study are those that are prisoners, under 18 years of age, or pregnant women.

Inclusion Criteria (Healthy Control Cohort):

* Staff in the enrolling site

Exclusion Criteria (Healthy Control Cohort):

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient Cohort: Patients admitted with a neurological or neurosurgical diagnosis that place them at risk for cerebral edema.
  Healthy Cohort: Faculty/Staff who interact with patients at the enrolling site
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Pupil's reaction to light as measured by Neurological Pupil Index (NPI) | 1 year
  Pupil's reaction to light as measured by Neurological Pupil Index (NPI) algorithm using pupillometer device that grades the pupil's reaction to light on a scale between 0 and 5. The Inter-device reliability is assessed using Cohen's Kappa method: values ≤ 0 as indicating no agreement.

CONTACTS AND LOCATIONS:
Overall Officials: DaiWai M Olson, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Clements University Hospital, Dallas, Texas, United States